CLINICAL TRIAL: NCT03522428
Title: Vitamin B12 Supplementation in Addition to Folic Acid and Iron Improves Hematological and Biochemical Markers in Pregnancy: a Randomized Controlled Trial
Brief Title: Vitamin B12 Pregnancy Supplementation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mirela Zec (Other)
Responsible Party: Sponsor-Investigator, Mirela Zec, master of laboratory medicine diagnostics, University of Split, School of Medicine
Organization: University of Split, School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: dupin
Record Dates: First submitted 2018-04-06; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy Anemia
Keywords: vitamin b12; pregnancy; anemia
MeSH Terms: conditions — Anemia | interventions — Vitamin B 12

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Receiving treatment (Active Comparator): Adding vitamin B12 at a dose of 5 μg / 100 days, custom folic acid therapy and iron supplements
  Interventions: Dietary Supplement: vitamin b12
- Control group (No Intervention): Standard prenatal care (custom folic acid therapy and iron supplements)

INTERVENTIONS:
Dietary Supplement: vitamin b12 — Vitamin B12 has been added to the experimental group of pregnant women, at a dose of 5 μg / 100 days
  Arms: Receiving treatment

SUMMARY:
Pregnancy is associated with increased requirements for iron and increased blood volume of up to 40%. Because expansion in plasma volume is higher than the increase in the mass of red blood cells, there is a fall in hemoglobin concentration, which leads to physiological anemia, characterized with lower hemoglobin (Hb), hematocrit and red blood cells, but without changes in mean corpuscular volume (MCV). Anemia in pregnancy is defined with Hb values under 110 g/L in the first trimester and under 105 g/L in the second and third trimester.

Iron deficiency is thought to be the most common nutrient deficiency among pregnant women. Consequences of anemia include delayed fetal growth, premature delivery, intrauterine fetal death, postpartum depression and delayed psychomotor development of a child. It is known that in women that are not anemic daily iron supplementation of 27 mg/day is sufficient, which can be obtained from adequate nutrition or body supplies. Iron supplementation is pregnancy has been recommended by the WHO (World Health Organisation) since 1959, and this recommendation was confirmed by numerous professional associations. However, in women with anemia, or women subjected to particular dietary regimens with diminished quantity of iron, including vegetarian or vegan diet, required supplementation dosage is higher, and estimated in the literature to be 120 mg/day.

The aim of this study was to analyze whether adding vitamin B12 (5 µg /100 days), along with folic acid and iron as supplement in pregnant women who are not anemic and who need only iron supplementation, will result in improvements of hematological and biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

* healthy women from 8th week of pregnancy

Exclusion Criteria:

* existence of hypertension
* existence of diabetes
* existence of genetic abnormalities
* smoking
* previous miscarriage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2012-12-23 (Actual); Study Completion 2012-12-23 (Actual)

PRIMARY OUTCOMES:
Change of Red blood cells (RBC) count in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  RBC count measured in SI (Systeme International) units (Nx10*12/L)
Change of Hemoglobin (Hgb) concentration in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  Hgb concentration in SI units (g/L)
Change of Hematocrit in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  volume percentage (%)
Change of Mean corpuscular volume (MCV) in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  mean volume of red blood cells in SI units (fL)
Change of Mean corpuscular hemoglobin concentration (MCHC) in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  Average hemoglobin concentration in a given volume of packed RBCs i SI units (g/L)
Change of Mean corpuscular hemoglobin (MCH) in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  average weight of hemoglobin in an average red blood cell in SI units (pg)
Change of Iron (Fe) in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  non-heme iron in serum in SI units (µmol/L)
Change of Haptoglobin in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  concentration of free haptoglobin in serum in SI units (g/L)
Change of Ferritin in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  serum ferritin in SI units (µg/L)
Change of Total Iron Binding Capacity (TIBC) in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  total iron binding capacity in SI units (µmol/L)
Change of Unsaturated Iron Binding Capacity (UIBC) in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  unsaturated iron binding capacity in SI units (µmol/L)

SECONDARY OUTCOMES:
Change of White Blood Cells (WBC) in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  RBC count measured in SI units (Nx10*9/L)
Change of Platelet Count in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  RBC count measured in SI units (Nx10*9/L)
Change of Transferrin in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  transferrin serum concentration in SI units (g/L)
Change of Neutrophils in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  proportion of neutrophils of all white cells (%)
Change of Lymphocytes in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  proportion of lymphocytes of all white cells (%)
Change of Monocytes in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  proportion of monocytes of all white cells (%)
Change of Eosinophils in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  proportion of eosinophils of all white cells (%)
Change of Basophils in first and second trimester | at two time points: on the 8th-10th and 22nd-24th weeks of pregnancy
  proportion of basophils of all white cells (%)

CONTACTS AND LOCATIONS:
Overall Officials: Damir Roje, Prof., Study Director — Clinical Hospital Center, Split